CLINICAL TRIAL: NCT04025463
Title: Enhancing Patient and Organizational Readiness for CVD Risk Reduction Among Persons Living With HIV or AIDS
Brief Title: Healing Our Hearts Minds and Bodies: CVD Reduction in Persons With HIV
Acronym: HHMB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Arleen F. Brown, MD, PhD, Principal Investigator, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1U01HL142109 (NIH); 1U01HL142109 (NIH)
Record Dates: First submitted 2019-06-27; First posted 2019-07-19 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: HIV/AIDS; Cardiovascular Risk Factors; Trauma, Psychological
Keywords: Implementation science; Organizational readiness; African American; Latino
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Psychological Trauma

STUDY DESIGN:
Intervention Model Description: Hybrid type II effectiveness/implementation study design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): Hybrid type II effectiveness/implementation study design - pre-post design with each participant serving as his or her own control.
  Interventions: Behavioral: HHMB

INTERVENTIONS:
Behavioral: HHMB — Blended, culturally-congruent, evidence-informed care model to increase patient and clinic participation in CVD risk reduction for patients with HIV

SUMMARY:
"Healing our Minds and Bodies" (HHMB) uses a a hybrid type II effectiveness/implementation study design to increase both patient and organizational readiness to address trauma and CVD risk among African American and Latino persons living with HIV or AIDS (PLWHIV).

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) has emerged as an increasingly important cause of morbidity and mortality among people living with HIV (PLWHIV). Now that HIV is considered a manageable chronic disease, the identification and treatment of comorbid medical conditions including CVD are increasingly the focus of research and clinical attention. What is missing, however, is yet another critical component of care for PLWHIV: integrated care for histories of trauma. Experiences of trauma increase the likelihood of HIV infection as well as CVD risk, yet health care for PLWHIV is rarely coordinated to address these three intersecting issues of HIV, CVD, and trauma, particularly among those disproportionately affected by HIV, i.e., ethnic minority patients. Histories of trauma among PLWHIV are associated with inconsistent treatment adherence and non-adherence, and trauma history alone is associated with poor CVD outcomes. Failure to address trauma poses significant barriers to the adoption of CVD risk strategies among PLWHIV. Health systems that coordinate and integrate care across HIV and chronic conditions such as CVD may provide the infrastructure needed to address the complex interplay of these conditions and their therapies. The investigators have designed a novel blended, culturally-congruent, evidence-informed care model, "Healing our Minds and Bodies" (HHMB), to address patients' trauma histories and barriers to care, and to prepare patients to engage in CVD risk reduction. Recognizing the need to ensure that PLWHIV receive CVD guideline-concordant care, the investigators have also identified implementation strategies to prepare providers and clinics for addressing CVD risk among their HIV-positive patients. Therefore, using a hybrid type II effectiveness/implementation study design, the goal of this study is to increase both patient and organizational readiness to address trauma and CVD risk among PLWHIV. The Specific Aims are: (1) to assess and enhance organizational readiness for addressing trauma and CVD risk among ethnic minority PLWHIV; specifically, a phased approach will drive the use of implementation strategies designed to educate, monitor, and support providers and staff in adhering to CVD care guidelines; (2) using mixed methods, to (a) evaluate the use and effectiveness of implementation strategies over time, and (b) identify barriers and facilitators to organizational adoption of guidelines, provider adherence to guidelines, feasibility, and sustainability; and (3) To evaluate the effect of HHMB on cognitive-behavioral, emotional, and clinical outcomes among 260 African American and Latino PLWHIV. The investigators will use the Replicating Effective Programs (REP) framework to guide the use of implementation strategies and the tailoring of the HHMB intervention within our participating implementation settings, and the Consolidated Framework for Implementation Research to guide the evaluation analyses.

ELIGIBILITY:
Organizational/Staff Eligibility

* Inclusion Criteria: staff employed by the participating agencies
* Exclusion Criteria: non-employees of the participating agencies

Patient Eligibility

* Inclusion Criteria

  * African American and Latino
  * Patient cared for in a participating agency
  * 18 to 60 years of age
  * Living with HIV or AIDS
  * Speak English or Spanish
  * Screen greater than 0 on the UCLA Life Adversities Screener (LADS)
  * Identify at least one self-reported CVD risk factor
* Exclusion Criteria - Potential participants will be screened by the Project Coordinator, who will be trained to assess the following exclusion criteria:

  * Known psychiatric, physical or neurological impairment that would limit their effective participation;
  * Recent history of a severe illness, sexual or physical abuse that might require sudden medical, psychological and/or legal intervention
  * Unwilling or unable to give consent or to commit to participate in the study through completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Experience of workload | Baseline
  Maslach Burnout Inventory - 16-item general survey measuring burnout in the workplace. Scale ranges from 0-6,with 0 = "Never" and 6 = "every day."
Implementation Climate Scale | Baseline
  This 18-item measure assesses the degree to which there is a strategic organizational climate supportive of evidence-based practice implementation. Implementation climate is defined as employees' shared perceptions of the policies, practices, procedures, and behaviors that are rewarded, supported, and expected in order to facilitate effective EBP implementation. The scale ranges from 0-4, with 0 = "not at all" and 4 = "very great extent."
Implementation Leadership Scale | Baseline
  The ILS assesses the degree to which a leader is Proactive, Knowledgeable, Supportive, and Perseverant in implementing evidence-based practice. The score for each subscale is created by computing a mean score for each set of items that load on a given subscale. For example, items 1, 2, and 3 constitute Scale 1. A mean of the scale scores may be computed to yield the mean score for the total ILS.
Implementation Citizenship Behavior Scale | Baseline
  This measure assesses the behaviors employees perform that exceed their expected job tasks to support the implementation of evidence-based practices (EBPs). The score for each subscale is created by computing a mean score for each set of items that load on a given subscale. For example, items 1, 2, and 3 constitute Scale 1 (Helping Others). A mean of the scale scores may be computed to yield the mean score for the total ICBS.
Change from baseline in CVD Risk - Life's Simple Seven | Three-month Follow-up
  Seven risk factors that individuals can improve through lifestyle changes to help achieve ideal cardiovascular health
Change from baseline in PROMIS V1.2 - Global Health | Three-month Follow-up
  Assessment of generic (not condition-specific) physical, mental, and social health. The adult PROMIS Global Health measure produces two scores: Physical Health and Mental Health.
Change from baseline in Difficulties in Emotional Regulation (DERS) | Three-month Follow-up
  Self-report measure of six facets of emotion regulation. Items are rated on a scale of 1 ("almost never [0-10%]") to 5 ("almost always [91-100%]"). Higher scores indicate more difficulty in emotion regulation.
Change from baseline in Woke Scale | Three-month Follow-up
  Measure of Critical Racial Consciousness

SECONDARY OUTCOMES:
Change from baseline in Hill-Bone Adherence Scale | Three-month Follow-up
  Medication adherence for medications for hypertension, diabetes, or hyperlipidemia
Change from baseline in HIV Adherence Scale | Three-month Follow-up
  Self-reported Rating, Frequency,
Change from baseline in Beck Depression Inventory-II | Three-month Follow-up
  Depression screener
Change from baseline in Overall Anxiety Severity and Impairment Scale (OASIS) | Three-month Follow-up
  Anxiety screener - 5-item
Change from baseline in Post-traumatic Stress (PDS-5) | Three-month Follow-up
  Estimates the severity of a respondent's PTSD symptoms.
Change from baseline in AUDIT-C | Three-month Follow-up
  Brief alcohol screen to identify hazardous drinking or active alcohol use disorders
Change from baseline in CAGE-AID | Three-month Follow-up
  Brief screen for alcohol and drug problems conjointly
Change from baseline in Pittsburgh Sleep Quality Index (PSQI) | Three-month Follow-up
  Measure of quality and patter of sleep in adults
Change from baseline in ASCVD Risk Score | Three-month Follow-up
  Estimate of 10-year and lifetime risks for atherosclerotic cardiovascular disease (ASCVD), defined as coronary death or nonfatal myocardial infarction, or fatal or nonfatal stroke. Sensitivity analyses will be conducted including and excluding those on a statin.

CONTACTS AND LOCATIONS:
Overall Officials: Gail Wyatt, PhD, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - OASIS Clinic, Los Angeles, California
  - Northeast Valley Healthcare Corporation, Van Nuys, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wyatt GE, Loeb TB, Cooley-Strickland M, Chin D, Wyatt LE, Smith-Clapham AM. Novel methodologies using history to document the effects of African American sexual trauma: Perspectives of Gail E. Wyatt, PhD. Am Psychol. 2023 May-Jun;78(4):563-575. doi: 10.1037/amp0001132. PMID 37384508
- [Background] Loeb TB, Viducich I, Smith-Clapham AM, Adkins-Jackson P, Zhang M, Cooley-Strickland M, Davis T, Pemberton JV, Wyatt GE. Unmet need for mental health services utilization among under-resourced Black and Latinx adults. Fam Syst Health. 2023 Jun;41(2):149-159. doi: 10.1037/fsh0000750. Epub 2022 Dec 15. PMID 36521110
- [Background] Loeb TB, Banks D, Ramm K, Viducich I, Beasley Q, Barron J, Chen EL, Norwood-Scott E, Fuentes K, Zhang M, Brown AF, Wyatt GE, Hamilton AB. Achieving Health Equity and Continuity of Care for Black and Latinx People Living With HIV. Am J Public Health. 2023 Jun;113(S2):S107-S109. doi: 10.2105/AJPH.2023.307222. No abstract available. PMID 37339419
- [Derived] Hamilton AB, Brown A, Loeb T, Chin D, Grills C, Cooley-Strickland M, Liu HH, Wyatt GE. Enhancing patient and organizational readiness for cardiovascular risk reduction among Black and Latinx patients living with HIV: Study protocol. Prog Cardiovasc Dis. 2020 Mar-Apr;63(2):101-108. doi: 10.1016/j.pcad.2020.02.014. Epub 2020 Feb 25. PMID 32109483

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-08): https://cdn.clinicaltrials.gov/large-docs/63/NCT04025463/Prot_SAP_000.pdf